CLINICAL TRIAL: NCT01956474
Title: Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas
Brief Title: CXL-04 A Study of Collagen Crosslinking With Ultraviolet-A in Asymmetric Corneas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXL-04
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Keratoconus
Keywords: keratoconus; cross-linking; Post-LASIK ectasia; Pellucid marginal degeneration; Forme fruste pellucid marginal degeneration; FFKC; Radial Keratotomy; Terrien's Marginal Degeneration
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Theralight crosslinking and Riboflavin (Other): ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) using UVA light and the photo- mediator riboflavin
  Interventions: Other: Theralight crosslinking and Riboflavin

INTERVENTIONS:
Other: Theralight crosslinking and Riboflavin — Corneal Collagen cross linking with UV light and riboflavin

SUMMARY:
The purpose of this study is to evaluate the efficacy of ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) as a method to increase the biomechanical and biochemical stability of the cornea by inducing additional cross-links within or between collagen fibers using UVA light and the photo- mediator riboflavin.

DETAILED DESCRIPTION:
This study will evaluate the results of Corneal Collagen Crosslinking (CXL) in patients with conditions that include Keratoconus, Pellucid Marginal degeneration, Post-LASIK ectasia, and patients with radial keratotomy who experience fluctuation in their vision. This is an outcomes study, all patients receive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 8 years of age or older
2. Having at least one of the following conditions:

   * Keratoconus
   * Post-LASIK ectasia
   * Pellucid marginal degeneration
   * Forme fruste pellucid marginal degeneration
   * FFKC
   * History of Radial Keratotomy with fluctuating vision.
   * Terrien's Marginal Degeneration
3. Signed written informed consent and/or assent
4. Likely to complete all study visits
5. Minimum corneal thickness of at least 250 microns measured by ultrasound or Pentacam for all indications other than Terrien's. For Terrien's, the minimal corneal thickness should be consistent with the surgeon's best surgical judgment.

Exclusion Criteria:

1. Severe corneal scarring that markedly affects vision
2. Contraindications to any study medications or their components
3. Pregnancy or breast feeding
4. Active Herpes Corneal Disease

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1324 (Actual)
Dates: Start 2013-01; Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Change in Best Spectacle Corrected Visual Acuity (BSCVA) | 6-9 months

SECONDARY OUTCOMES:
Change in Uncorrected Visual Acuity (UCVA) | 6-9 months
Change in Corneal topography | 6-9 months
Change in Manifest Refraction | 6-9 months
Change in Keratometry on topography and Pentacam | 6-9 months
Change in Wavefront Refraction and aberrations | 6-9 months

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — Cxlusa
Locations (6):
- United States (6):
  - Center for Excellence in Eye Care, Miami, Florida
  - Stulting Research Center at Woolfson Eye Institute, Atlanta, Georgia
  - TLC Laser Eye Center, Rockville, Maryland
  - Talamo Hatch Laser Eye Consultants, LLC, Boston, Massachusetts
  - Cleveland Eye Clinic, Brecksville, Ohio
  - TLC Laser Eye Center, Fairfax, Virginia